CLINICAL TRIAL: NCT07182565
Title: A Phase Ib/II Study of Hypofractionated Radiotherapy Combined With Immunochemotherapy as Neoadjuvant Treatment for Adenocarcinoma of the Gastroesophageal Junction
Brief Title: Hypofractionated Radiotherapy Plus Immunochemotherapy for Neoadjuvant Treatment of Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yaqin Zhao, Associate Chief Physician, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEJA-nICRT-2025-05
Record Dates: First submitted 2025-07-09; First posted 2025-09-19 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-07

CONDITIONS: Gastroesophageal Junction Adenocarcinoma; Hypofractionated Radiotherapy
Keywords: neoadjuvant therapy; hypofractionated radiotherapy; immunotherapy; chemotherapy; Serplulimab; pCR
MeSH Terms: interventions — Radiation Dose Hypofractionation; Immune Checkpoint Inhibitors; titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (HFRT+nICT) (Experimental)
  Interventions: Radiation: hypofractionated radiotherapy; Drug: PD-1 inhibitor; Drug: TS-1
- Control Arm (nICT) (Active Comparator)
  Interventions: Drug: PD-1 inhibitor; Drug: TS-1

INTERVENTIONS:
Radiation: hypofractionated radiotherapy — In Phase Ib, hypofractionated radiotherapy (HFRT) will be administered at one of three dose levels: 3 Gy × 5 fractions, 4 Gy × 5 fractions, or 5 Gy × 5 fractions. The recommended dose determined in Phase Ib will be used in Phase II (delivered as 5 fractions).
  Other Names: HFRT; LFRT
  Arms: Intervention Arm (HFRT+nICT)
Drug: PD-1 inhibitor — Serplulimab will be administered concurrently with chemotherapy at a fixed dose of 300 mg via intravenous infusion on Day 1 of each 3-week cycle.
Drug: TS-1 — The TS regimen includes paclitaxel at a dose of 175 mg/m² administered via intravenous infusion on Day 1, and oral administration of tegafur-gimeracil-oteracil (S-1) for 14 consecutive days followed by a 7-day rest period (21-day cycle). The S-1 dose is based on body surface area (BSA): 40 mg twice daily (bid) for BSA ≤ 1.5 m²; 50 mg bid for BSA 1.5-1.6 m²; and 60 mg bid for BSA ≥ 1.6 m².

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of HFRT plus neoadjuvant ICT in locally advanced resectable GEJA.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether hypofractionated radiotherapy combined with a PD-1 inhibitor (Serplulimab) and chemotherapy based on the TS regimen is a safe and well-tolerated neoadjuvant strategy for patients with locally advanced resectable gastroesophageal junction adenocarcinoma (GEJA), and whether it can improve the pathological complete response (pCR) rate compared to immunochemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed diagnosis of locally advanced adenocarcinoma of the gastroesophageal junction (GEJ) (Siewert types I-III), defined as cT3-4, any N, M0 or cT2 N+, M0 according to the 8th edition of the AJCC staging system.
2. Determined as resectable locally advanced disease after multidisciplinary team (MDT) evaluation.
3. Age ≥18 years, regardless of sex.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
5. Estimated life expectancy ≥3 months.
6. No prior anti-cancer treatment.
7. At least one measurable lesion as defined by RECIST v1.1 (lesion diameter ≥1 cm on spiral CT or ≥2 cm on standard CT or MRI), assessed within 28 days prior to enrollment.
8. Adequate organ function within 14 days prior to treatment, defined as follows (note: blood transfusions, platelet infusions, or G-CSF use not permitted within 14 days prior to hematologic assessment):

1) Hematological: Hemoglobin ≥9 g/dL (without recent transfusion); ANC ≥1.5 × 10⁹/L; WBC ≥3.0 × 10⁹/L (no G-CSF use); Platelets ≥75 × 10⁹/L (no IL-11 or TPO use).

2) Biochemistry: Total bilirubin ≤1.5 × ULN; AST and ALT ≤2.5 × ULN; Serum creatinine ≤1.5 × ULN or creatinine clearance ≥60 mL/min (Cockcroft-Gault formula); Serum albumin ≥25 g/L.

3) Coagulation: INR <1.5, APTT <1.5 × ULN within 7 days before enrollment; PT ≤1.5 × ULN.

9.Patients with active hepatitis B or C infection must have received antiviral therapy ≥14 days prior to enrollment, with HBV DNA ≤500 IU/mL or 2500 copies/mL, HCV RNA undetectable, and agree to continue antiviral therapy during the study.

10.LVEF ≥50% on echocardiography. 11.Women of childbearing potential must have a negative pregnancy test (serum or urine) within 7 days prior to enrollment and agree to use effective contraception during the study and for at least 3 months after the last dose. Males must use effective contraception during and for at least 3 months after treatment. Female participants must not be breastfeeding or donate/retrieve ova within 60 days after the last dose.

12.Willing and able to provide written informed consent and comply with study procedures.

Exclusion Criteria:

1. Confirmed dMMR or MSI-H by immunohistochemistry or genetic testing.
2. Evidence of peritoneal or visceral metastasis (based on thoracoabdominal CT, bone scan, or MRI if bone metastasis is suspected).
3. Other malignancies within the past 5 years, except cured basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix.
4. Known allergy or hypersensitivity to any study drugs or their excipients; contraindications to study drugs.
5. Clinically significant upper gastrointestinal bleeding within 30 days before enrollment or randomization.
6. Interstitial lung disease, pulmonary fibrosis, active tuberculosis, or steroid-requiring pneumonitis confirmed by CT.
7. Active autoimmune or inflammatory disease requiring immunosuppressants within 2 years (e.g., IBD, SLE, sarcoidosis, Wegener's, MG, Graves', rheumatoid arthritis, etc.); exceptions: well-controlled type 1 diabetes, hypothyroidism under hormone replacement, untreated localized skin diseases (e.g., vitiligo, psoriasis).
8. Immunodeficiency, history of HIV infection or organ transplantation.
9. Active HBV (HBsAg positive) or HCV infection. Previously treated or well-controlled HBV/HCV is allowed.
10. Systemic corticosteroids or immunosuppressants within 2 weeks prior to treatment. Exceptions: inhaled or local steroids, adrenal replacement (<10 mg/day prednisone equivalent), or short-term corticosteroids (<7 days) for prophylaxis or non-autoimmune indications.
11. Uncontrolled comorbidities, including:

1）Poorly controlled hypertension (SBP ≥150 mmHg or DBP ≥100 mmHg); 2）Grade II+ myocardial ischemia or MI within 6 months, arrhythmia (QT ≥480 ms, AF), uncontrolled angina, CHF (NYHA III-IV), valvular disease, cardiomyopathy, stroke or TIA history; 3）Active or uncontrolled infection; 4）Liver disease (cirrhosis, decompensation, active hepatitis); 5）Poorly controlled diabetes (FBG >10 mmol/L); 6）Proteinuria ≥++ or 24h urine protein >1.0 g. 12.Coagulation abnormalities (INR >1.5 or APTT >1.5 × ULN), known bleeding tendency, or patients receiving thrombolytic or anticoagulant therapy. Known congenital or acquired bleeding or thrombotic disorders, such as hemophilia, coagulation defects, thrombocytopenia, hypersplenism, etc.

Patients with significant hemoptysis (≥2.5 mL per day), or a history of clinically significant bleeding (e.g., gastrointestinal bleeding, hemorrhagic gastric ulcers, or fecal occult blood test ≥++) within 3 months prior to enrollment.

Patients requiring long-term anticoagulation with warfarin or heparin, or long-term antiplatelet therapy (aspirin ≥300 mg/day or clopidogrel ≥75 mg/day).

13.Major surgery (e.g., craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to first dose, or expected to undergo major surgery during the study, or non-diagnostic surgery within 4 weeks prior to trial initiation.

14.History of gastrointestinal perforation and/or fistula within 6 months before enrollment; or history of arterial or venous thromboembolic events, such as stroke (except stable cerebral infarction as judged by the investigator), deep vein thrombosis, or pulmonary embolism.

15.Long-term unhealed wounds or fractures. 16.Severe gastrointestinal conditions that may interfere with oral drug absorption, such as inability to swallow, chronic diarrhea, or intestinal obstruction.

17.Severe malnutrition. 18.Pregnant or lactating women, or participants of reproductive potential (male or female not postmenopausal for at least one year) who are unwilling to use effective contraception.

19.History of substance abuse or uncontrolled psychiatric illness. 20.Unwillingness or inability to comply with study requirements. 21.Participation in another clinical trial within 30 days prior to study entry, or planning to participate in another trial during the study period.

22.Any severe or uncontrolled medical condition, judged by the investigator to potentially compromise patient safety or interfere with study completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability in Phase Ib | within 3 months after the HFRT
  Safety will be assessed based on clinical adverse events, vital signs, and abnormalities in laboratory tests during the study period.
  Adverse events (AEs) will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
  All deaths occurring within 90 days after the first dose of treatment or within 30 days after the last dose will be listed along with the causes of death.
  Laboratory abnormalities will be categorized according to NCI-CTCAE version 5.0.
  Maximum Tolerated Dose (MTD): If ≥1/3 of patients in a given dose cohort experience radiotherapy-related dose-limiting toxicities (DLTs) within 90 days, that dose level will be considered intolerable. The dose level immediately below will then be defined as the maximum tolerated dose (MTD). At least six evaluable patients are required in the MTD cohort.
pCR rate in Phase II | approximately 2 weeks after the resection of primary lesion
  pCR rate: The proportion of patients who achieve pathological complete response (pCR), defined as the absence of viable tumor cells on microscopic examination after neoadjuvant therapy.

SECONDARY OUTCOMES:
R0 resection rate | approximately 2 weeks after the resection of primary lesion
  number of R0 surgery divide all participants
Objective response rate | From Baseline up to the pre-surgical assessment (performed within 28 days after the last dose of conversion therapy)
  Objective response rate (ORR) is defined as the proportion of subjects with a confirmed Complete Response (CR) or Partial Response (PR) as assessed by the investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. A response (CR or PR) requires confirmation by a repeat assessment performed no less than 4 weeks after the criteria for response are first met.
DFS(disease free survival) rate | Up to 3 years
  evaluate the DFS rate after the resection of primary lesion（only patients who acquire R0 resection）
OS(overall survival) rate | Up to 3 years
  evaluate the OS rate after the neoadjuvant therapy
Adverse Events (AEs) | From the first dose through 90 days after the last dose
  The incidence, severity, and relationship of adverse events will be assessed and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0.
Quality of Life (QoL) - EORTC QLQ-C30 | Assessments are performed at Baseline, on Day 1 of each subsequent treatment cycle (each cycle is 21 days), at the end-of-treatment visit, and at 1, 3, 6, and 12 months post-surgery during follow-up.
  Quality of life will be evaluated using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30).

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - West China Xiamen Hospital, Sichuan University, Xiamen, Fujian
  - The Seventh People's Hospital of Chengdu, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - West China Shangjin Nanfu Hospital, Sichuan University, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Yes
IPD(individual patient data) Sharing Plan: Shared for: scientific research institutions, academic journal editors, government agencies Sharing conditions: IPD sharing shall meet the following conditions: Requestor must provide study agreement and relevant ethical review committee approval documents Requestor must ensure legality of data use and privacy protection Requestor must agree to data sharing, and the study team has the right to review the Requestor 's study plan and provide necessary support and interpretation of data
  Scope of shared data: The shared data includes ECG and clinical data of all subjects, but excluding personal information of subjects
Time Frame: Sharing period is 5 years, which start from one year after primary outcome publication.
Access Criteria: Shared for: scientific research institutions, academic journal editors, government agencies Sharing conditions: IPD sharing shall meet the following conditions: Requestor must provide study agreement and relevant ethical review committee approval documents Requestor must ensure legality of data use and privacy protection Requestor must agree to data sharing, and the study team has the right to review the Requestor 's study plan and provide necessary support and interpretation of data